CLINICAL TRIAL: NCT06519058
Title: Effectiveness of Carpal Ligament Self-Myofascial Stretching Over Conventional Physical Therapy on Reducing Pain and Improving Function in Patients With Stage I and II Carpal Tunnel Syndrome
Brief Title: Effectiveness of Self-Myofascial Stretching on Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Shibili Nuhmani, Assistant professor, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: (AWH/EC/01/2022)
Record Dates: First submitted 2024-06-27; First posted 2024-07-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Patients With Stage I and II Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- self-myofascial stretching group (Experimental)
  Interventions: Other: self-myofascial stretching
- conventional physical therapy group (Sham Comparator)
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Other: self-myofascial stretching — self-myofascial stretching exercise
  Arms: self-myofascial stretching group
Other: conventional physical therapy — conventional physical therapy treatment, including exercises
  Arms: conventional physical therapy group

SUMMARY:
Background/Objectives: Carpal tunnel syndrome (CTS), a median mononeuropathy from nerve compression in the wrist's carpal tunnel, will be studied to compare self-myofascial carpal ligament stretching plus conventional physical therapy versus physical therapy alone for pain reduction and function improvement in stage I/II CTS patients.

Methods: Thirty-six eligible stage I/II CTS patients will be randomized (18/group). The experimental group will receive self-myofascial stretching + conventional therapy; controls will get conventional therapy only. Treatment will last 6 weeks; outcomes will be assessed via Boston Carpal Tunnel Questionnaire and Visual Analogue Scale.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed CTS, stage I/II (EMG-confirmed).

Age 30-60 years.

Both genders.

Dominant hand (unilateral/bilateral).

English literate.

Exclusion Criteria:

Polyneuropathy.

Adaptive equipment use.

Shoulder pathologies.

Other neurological/musculoskeletal conditions.

Recent carpal tunnel release (<1 year).

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-04 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Questionnaire | 6 weeks
  Used to assess the function of carpals
Visual Analogue Scale | 6 weeks
  Involves asking participants to rate their current level of pain on a scale from 0= No pain to 10= maximum pain is felt.

CONTACTS AND LOCATIONS:
Overall Officials: Shibili Nuhmani, PhD, Principal Investigator — Imam Abdulrahman Bin Faisal University
Locations (1):
- Awh special college, Calicut, India